CLINICAL TRIAL: NCT03328884
Title: Multicenter Open-label, Phase II Trial, to Evaluate the Efficacy and Safety of Nal-IRI for Progressing Brain Metastases in Patients With HER2-negative Breast Cancer (The Phenomenal Study)
Brief Title: Evaluation of the Efficacy and Safety of Nal-IRI for Progressing Brain Metastases in Breast Cancer Patients
Acronym: Phenomenal
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedSIR (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MedOPP107; 2016-002689-30 (EudraCT Number)
Record Dates: First submitted 2017-03-17; First posted 2017-11-01 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer Metastatic
MeSH Terms: interventions — Irinotecan; Liposomes; irinotecan sucrosofate

STUDY DESIGN:
Intervention Model Description: This is an international, prospective, open-label, multicenter, single arm, two-stage Simon Design phase II clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nal-IRI (Other): This is a single arm study. After signing the informed consent form, patients will start treatment with nal-IRI. nal-IRI will be administered 50 mg/m2 on D1 of a 14-day cycle in monotherapy.
  Interventions: Drug: Irinotecan (CPT-11) liposome

INTERVENTIONS:
Drug: Irinotecan (CPT-11) liposome — nal-IRI (nanoliposomal irinotecan, also known as MM-398 and PEP02) is irinotecan free base, (also known as CPT-11) a topoisomerase 1 inhibitor, encapsulated in a liposome drug delivery system.
  nal-IRI will be administered 50 mg/m2 on D1 of a 14-day cycle in monotherapy.
  Other Names: nal-IRI

SUMMARY:
Multicenter open-label, phase II trial, to evaluate the efficacy and safety of nal-IRI in patients with HER2-negative breast cancer, who have documented Central Nervous System (CNS) progression following Whole Brain Radio Therapy (WBRT), Stereotactic Radiosurgery (SRS) and/or surgery, as determined by the Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM) criteria.

DETAILED DESCRIPTION:
This is an international, prospective, open-label, multicenter, single arm, two-stage Simon Design phase II clinical trial, with the primary objective of assessing the efficacy of nal-IRI single agent in a cohort of HER2-negative metastatic breast cancer (MBC) patients with CNS involvement.

Eligible patients will have histologically proven diagnosis of adenocarcinoma of the breast, they must have progressed to at least one prior chemotherapy regimen in the metastatic setting and must have been progressed in CNS to previous local treatment (Surgery and/or WBRT and/or SRS) showing at least one measurable lesion in the CNS (symptomatic meningeal carcinomatosis is not permitted). Eligible patients must have been previously received at least treatment with taxanes (either in the neo/adjuvant or in the metastatic scenario). Patients could not be eligible if they are candidates for a local treatment with a radical intention.

Patients will be accrued in a two-stage design. Considering a drop-out rate of 10%, the accrual goal will be a total of 63 patients in both stages (first stage will include 23 evaluable patients and the second stage will include 33 more evaluable patients).

ELIGIBILITY:
Inclusion Criteria:

1. Female or male patients > 18 years
2. Patients must have a diagnosis of metastatic breast cancer.
3. Patients should have been pretreated with taxanes at any time prior to the study enrolment if not formally contraindicated.
4. At least one prior chemotherapy regimen for advanced disease.
5. Evidence of new brain metastases and/or stable or progressive brain metastases following previous WBRT and/or SRS and/or surgery.
6. At least one brain lesion needed to be measurable for new and progressive metastases (≥10 mm on T1-weighted, gadolinium-enhanced magnetic resonance imaging). For stable brain metastases at least one extracerebral lesion need to be measurable.
7. HER2 negative breast cancer defined as 0 - 1+ by immunohistochemistry or FISH negative result.
8. ECOG performance status <2.
9. Life expectancy >12 weeks.
10. Patients must have sufficient organ and marrow function as defined below:

    a. Hematopoietic parameters: i. Absolute neutrophil count ≥ 1,5 x 109/L ii. Platelets ≥ 100 x 109/L iii. Haemoglobin ≥ 9 mg/dL b. Hepatic parameters: i. Total bilirubin ≤ 1.5 mg/dL ii. AST (SGOT)/ALT (SGPT) ≤ 2.5 X institutional upper limit of normal c. Renal parameters: i. Creatinine ≤ 1.5 X institutional upper limits of normal, OR ii. Creatinine clearance ≥ 60 mL/min/1.73 m2 for pts w/ creatinine levels > institutional normal.
11. Participants of childbearing potential must agree to use at least efficient contraception method (even though it is recommendable for them to use a highly effective method) prior to study entry and for the duration of study participation as well as a negative serum pregnancy test within 7 days of study enrolment and at the end of treatment visit.
12. Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

1. Patients must not have previously received nal-IRI or any other form of irinotecan, conventional or liposomal.
2. Patients who have received prior anti-cancer treatment with chemotherapy, endocrine therapy, immunotherapy or radiotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin-C) prior to starting study treatment.
3. Radiation therapy encompassing more than 30% of bone marrow.
4. Significant chronic gastrointestinal disorder with diarrhea as a major symptom (i.e Crohn's disease, ulcerative colitis, malabsorption, or grade ≥ 2 diarrhea of any etiology at baseline)
5. Have a serious concomitant systemic disorder (e.g. active infection including HIV, or cardiac disease) incompatible with the study (at the discretion of investigator), previous history of bleeding diathesis, or treatment with Sintrom.
6. Patients who have symptomatic lymphangitis, dyspnoea at rest or meningeal carcinomatosis. (Patients with asymptomatic involvement may be enrolled in the study.)
7. Patients must be recovered from any clinically relevant toxic effects of any prior surgery, radiotherapy or other therapy intended for the treatment of breast cancer. For peripheral neuropathy, up to CTCAE (v4.0) Grade 2 is acceptable for patients with pre-existing condition.
8. Patients may not be receiving any other investigational or anticancer agents while on the study.
9. History of other malignancies, which could affect compliance with the protocol or interpretation of the results. Patients with malignancies diagnosed more than 5 years prior to study day 1, adequately treated carcinoma in situ of the cervix or basal or squamous cell skin are generally eligible.
10. Pregnant or lactating women.
11. NYHA Class III or IV congestive heart failure, ventricular arrhythmias or uncontrolled blood pressure. Or known abnormal ECG with clinically significant abnormal findings.
12. Active infection or an unexplained fever >38.5°C (excluding tumoral fever), which in the physician's opinion might compromise the patient's health.
13. Patients with other significant disease or disorders that, in the Investigator's opinion, would exclude the patient from the study.
14. Current use or any use in the last two weeks of strong CYP3A-enzyme inducers/inhibitors and/or strong UGT1A inhibitors
15. Known hypersensitivity to any of the components of nanoliposomal irinotecan (nal-IRI) other liposomal irinotecan formulations or irinotecan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2025-04-02 (Actual)

PRIMARY OUTCOMES:
CNS Overall Response Rate (ORR) | From Baseline up to 80 weeks after patient entry
  The efficacy of nal-IRI will be measured in terms of CNS ORR, defined as per RANO-BM criteria. According to these criteria Complete Response (CR) will be defined as the disappearance of all CNS target lesions sustained for at least 4 weeks; no new lesions, no corticosteroids; stable or improved clinically. Partial Response (PR) will be defined as a decrease of at least 30% in the sum longest diameter (LD) of CNS target lesions, taking as reference the baseline sum LD, sustained for at least 4 weeks; no new lesions; no corticosteroids; stable or improved clinically.

SECONDARY OUTCOMES:
CNS disease stabilization on week 12 | From Baseline up to 12 weeks after patient entry
  CNS clinical benefit rate (CBR) at week 12 will be defined as the percentage of patients who experience a CR, PR or Stable Disease (SD) for at least 12 weeks assessed by the modified Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST v.1.1) criteria.
ORR, according to a volumetric parameter, and to the RECIST v.1.1 criteria | From Baseline up to 80 weeks after patient entry
  ORR according to a volumetric parameter. For this objective, PR will be defined as > 65% volumetric reduction of CNS lesion(s) and to the RECIST v.1.1 criteria. The volumetric parameter will be centrally reviewed.
CBR | 3 years
  The percentage of patients who experience a CR, PR or SD for at least 24 weeks and assessed by the RECIST v.1.1 criteria.
Safety profile of nal-IRI in this population by Common Terminology Criteria for Adverse Events version 4 (CTCAE v.4) criteria | 3 years
  This study will consider the National Cancer Institute (NCI) CTCAE v.4 criteria grade 3 and 4 adverse events (AEs) and serious AEs (SAEs) in order to assess the safety and tolerability objectives.
Progression-Free Survival (PFS) | 3 years
  PFS will be defined as the time from the first dose of treatment to death or disease progression as assessed by the Investigator per RECIST v1.1 criteria.
Overall Survival (OS) | 3 years
  OS will be defined as the time from the first dose of treatment to death for any cause.
Disease Control Rate | 18 months after last patient included
  DCR will be defined as the percentage of patients who experience a CR, PR or stable disease determined locally by the investigator, using RANO-BM criteria (for IC lesions) and RECIST criteria v.1.1 (for IC, EC, and overall lesions) in patients with progressing brain metastases and in all patients with CNS involvement.
TTR | From treatment initiation to time of the first objective tumor response in patients with CR or PR,
  TTR will be defined as the time from treatment initiation to time of the first objective tumor response observed in patients who achieved a CR or PR, determined locally by the investigator, using RANO-BM criteria (for IC lesions) and RECIST criteria v.1.1 (for IC, EC, and overall lesions) in patients with progressing brain metastases and in all patients with CNS involvement.
DoR | time from the first occurrence of a documented objective response to disease progression or death
  DoR will be defined as the time from the first occurrence of a documented objective response to disease progression or death from any cause, whichever occurs first, determined locally by the investigator, using RANO-BM criteria (for IC lesions) and RECIST criteria v.1.1 (for IC, EC, and overall lesions) in patients with progressing brain metastases and in all patients with CNS involvement.
MTS | From baseline
  MTS from baseline in the size of target tumor lesions, defined as the biggest decrease, or smallest increase if no decrease observed, determined locally by the investigator, using RANO-BM criteria (for IC lesions) and RECIST criteria v.1.1 (for IC, EC, and overall lesions) in patients with progressing brain metastases and in all patients with CNS involvement.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Cortes, Principal Investigator — Hospital Universitario Ramon y Cajal
Locations (16):
- Spain (16):
  - ICO, Badalona
  - IOB Institute of Oncology - Quirón Barcelona, Barcelona
  - Hospital Universitario Virgen de Las Nieves, Granada
  - Hospital Universitario Clinico San Cecilio, Granada
  - H. Ruber Juan Bravo, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Doce de Octubre, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - MD Anderson Madrid, Madrid
  - Hospital Clínico Virgen de la Victoria, Málaga
  - Hospital Universitari Son Espases, Palma de Mallorca
  - Son Llatzer, Palma de Mallorca
  - Sant Joan de Reus, Reus
  - Hospital Universitario Virgen del Rocío, Seville
  - IVO, Valencia
  - H. Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No
It is not planned